CLINICAL TRIAL: NCT03510715
Title: An Open-Label Study to Evaluate the Efficacy and Safety of Alirocumab in Children and Adolescents With Homozygous Familial Hypercholesterolemia
Brief Title: An Efficacy and Safety Study of Alirocumab in Children and Adolescents With Homozygous Familial Hypercholesterolemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EFC14660; 2017-002297-39 (EudraCT Number); U1111-1200-2046 (Other: UTN)
Record Dates: First submitted 2018-04-18; First posted 2018-04-27 (Actual); Results first posted 2020-12-29 (Actual); Last update posted 2020-12-29 (Actual); Status verified 2020-10

CONDITIONS: Hypercholesterolemia
Keywords: Pediatrics, Homozygous Familial Hypercholesterolemia, Alirocumab, PCSK9 inhibitor, Low-density Lipoprotein Cholesterol (LDL-C)
MeSH Terms: conditions — Hypercholesterolemia; Homozygous Familial Hypercholesterolemia | interventions — alirocumab; Atorvastatin; Simvastatin; Fluvastatin; Pravastatin; Lovastatin; Rosuvastatin Calcium; Ezetimibe; Cholestyramine Resin; Niacin; Fenofibrate; Fatty Acids, Omega-3

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Alirocumab (Experimental): Participants with BW less than (<) 50 kilograms (kg) received subcutaneous (SC) injection of alirocumab 75 mg Q2W for 48 weeks. Alirocumab dose was up-titrated to 150 mg Q2W from Week 12 in case of increase in BW with BW greater than or equal to [>=] 50 kg.
  Participants with BW >=50 kg received SC injection of alirocumab 150 mg Q2W for 48 weeks.
  Interventions: Drug: Alirocumab SAR236553 (REGN727); Drug: Atorvastatin; Drug: Simvastatin; Drug: Fluvastatin; Drug: Pravastatin; Drug: Lovastatin; Drug: Rosuvastatin; Drug: Ezetimibe; Drug: Cholestyramine; Drug: Nicotinic acid; Drug: Fenofibrate; Drug: Omega-3 fatty acids

INTERVENTIONS:
Drug: Alirocumab SAR236553 (REGN727) — Pharmaceutical form: solution for injection in pre-filled syringe,
  Route of administration: subcutaneous (SC)
Drug: Atorvastatin — Pharmaceutical form: tablet,
  Route of administration: oral
Drug: Simvastatin — Pharmaceutical form: tablet,
  Route of administration: oral
Drug: Fluvastatin — Pharmaceutical form: capsule,
  Route of administration: oral
Drug: Pravastatin — Pharmaceutical form: tablet,
  Route of administration: oral
Drug: Lovastatin — Pharmaceutical form: tablet,
  Route of administration: oral
Drug: Rosuvastatin — Pharmaceutical form: tablet,
  Route of administration: oral
Drug: Ezetimibe — Pharmaceutical form: tablet,
  Route of administration: oral
Drug: Cholestyramine — Pharmaceutical form: oral suspension,
  Route of administration: oral
Drug: Nicotinic acid — Pharmaceutical form: tablet,
  Route of administration: oral
Drug: Fenofibrate — Pharmaceutical form: tablet,
  Route of administration: oral
Drug: Omega-3 fatty acids — Pharmaceutical form: capsule,
  Route of administration: oral

SUMMARY:
Primary Objective:

To evaluate the efficacy of alirocumab (75 or 150 milligrams [mg] depending on body weight [BW]), administered every 2 weeks (Q2W), on low-density lipoprotein cholesterol (LDL-C) levels at Week 12 of treatment in children and adolescents with homozygous familial hypercholesterolemia (hoFH) of 8 to 17 years of age on top of background treatments.

Secondary Objectives:

* To evaluate the efficacy of alirocumab after 24 and 48 weeks of treatment on LDL-C levels.
* To evaluate the effects of alirocumab on other lipid parameters (eg, apolipoprotein B [Apo B], non-high density lipoprotein cholesterol [non-HDL-C], total cholesterol [Total-C], high density lipoprotein cholesterol [HDL-C], lipoprotein a [Lp (a)], triglycerides [TG], apolipoprotein A-1 [Apo A-1] levels) after 12, 24, and 48 weeks of treatment.
* To evaluate the safety and tolerability of alirocumab up to 48 weeks of treatment.

DETAILED DESCRIPTION:
The study duration was up to 62 weeks, which included (if needed) a run-in period of up to 4 weeks, a screening period of up to 2 weeks, a treatment period of up to 48 weeks, and a follow-up of 8 weeks.

ELIGIBILITY:
Inclusion criteria :

* Participants genetically diagnosed with hoFH.
* Participants treated with optimal dose of statin +/- other lipid modifying therapies (LMTs), or non-statin LMTs if statin-intolerant at stable dose(s) for at least 4 weeks.
* A signed informed consent indicating parental permission with or without participants assent.
* For participants on apheresis, currently undergoing stable LDL apheresis therapy prior to the screening visit (Week -2) and had initiated apheresis treatment for at least 6 months.

Exclusion criteria:

* Participants with LDL-C <130 milligram per deciliter [mg/dL] (3.37 millimoles per liter [mmol/L]) obtained during the screening period after the participant had been on stable apheresis procedure or LMT (i.e., stable optimal dose of statin ± other stable LMTs, or stable non statin LMTs in statin-intolerant participants) treatment for at least 4 weeks.
* Participants with BW <25 kg.
* Participants aged 8 to 9 years not at Tanner Stage 1 and participants aged of 10 to 17 years not at least at Tanner Stage 2 in their development.
* Participants with uncontrolled Type 1 or 2 diabetes mellitus.
* Participants with known uncontrolled thyroid disease.
* Participants with uncontrolled hypertension.
* Participants who will receive statin de novo during the run-in period.
* Fasting triglycerides greater than (>) 350 mg/dL (3.95 mmol/L) at the screening visit.
* Severe renal impairment (i.e., estimated glomerular filtration rate <30 milliliter per minute/1.73 meter square) at the screening visit.
* Alanine aminotransferase or aspartate aminotransferase >2 * upper limit of normal (ULN) at the screening visit.
* Creatine phosphokinase >3 * ULN at the screening visit.

The above information was not intended to contain all considerations relevant to a participants potential participation in a clinical trial.

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 18 (Actual)
Dates: Start 2018-08-31 (Actual); Primary Completion 2020-02-17 (Actual); Study Completion 2020-02-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (10):
- Investigational Site Number 0760001, São Paulo, Brazil
- Investigational Site Number 1240001, Québec, Canada
- Investigational Site Number 2080001, Viborg, Denmark
- Investigational Site Number 4840006, Oaxaca City, Mexico
- Investigational Site Number 5280001, Amsterdam, Netherlands
- Investigational Site Number 6430002, Kemerovo, Russia
- Investigational Site Number 7050001, Ljubljana, Slovenia
- Investigational Site Number 7240001, A Coruña, Spain
- Investigational Site Number 1580001, Taipei, Taiwan
- Investigational Site Number 7920001, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bruckert E, Caprio S, Wiegman A, Charng MJ, Zarate-Morales CA, Baccara-Dinet MT, Manvelian G, Ourliac A, Scemama M, Daniels SR. Efficacy and Safety of Alirocumab in Children and Adolescents With Homozygous Familial Hypercholesterolemia: Phase 3, Multinational Open-Label Study. Arterioscler Thromb Vasc Biol. 2022 Dec;42(12):1447-1457. doi: 10.1161/ATVBAHA.122.317793. Epub 2022 Nov 3. PMID 36325897

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 10 active centers (which screened at least 1 participant) in 10 countries worldwide. Overall, 20 participants were screened between 31 August 2018 and 4 January 2019, of whom 2 were screen failures. Of the 10 centers which screened participants, 9 centers enrolled at least 1 participant.
Pre-assignment Details: A total of 18 participants were enrolled and received treatment in this study.
Groups:
- Alirocumab 75 mg Q2W/up to 150 mg Q2W: Participants with body weight (BW) less than (<) 50 kilograms (kg) received subcutaneous (SC) injection of alirocumab 75 milligrams (mg) every 2 weeks (Q2W) for 48 weeks. Alirocumab dose was up-titrated to 150 mg Q2W from Week 12 in case of increase in BW with BW greater than or equal to [>=] 50 kg.
- Alirocumab 150 mg Q2W: Participants with BW >=50 kg received SC injection of alirocumab 150 mg Q2W for 48 weeks.
Period: Overall Study
Arm/Group | Alirocumab 75 mg Q2W/up to 150 mg Q2W | Alirocumab 150 mg Q2W
Started | 9 | 9
Completed | 8 | 9
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Population: Analysis was performed on all enrolled participants.
Groups:
- Alirocumab 75 mg Q2W/up to 150 mg Q2W: Participants with BW <50 kg received SC injection of alirocumab 75 mg Q2W for 48 weeks. Alirocumab dose was up-titrated to 150 mg Q2W from Week 12 in case of increase in BW with BW >=50 kg.
- Total: Total of all reporting groups
Arm/Group | Alirocumab 75 mg Q2W/up to 150 mg Q2W | Alirocumab 150 mg Q2W | Total
Number analyzed (Participants) | 9 | 9 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.4 (1.5) | 14.3 (2.4) | 12.4 (2.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 9
  Male | 5 | 4 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 3
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 6 | 5 | 11
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Low-Density Lipoprotein Cholesterol (LDL-C) [Mean (Standard Deviation); unit: milligrams per deciliter (mg/dL)] | 437.7 (192.8) | 308.3 (181.6) | 373.0 (193.5)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Low-Density Lipoprotein Cholesterol (LDL-C) at Week 12: Intent-to-Treat (ITT) Analysis
Description: Adjusted least square (LS) means and standard errors were obtained from the mixed model analysis with repeated measures (MMRM) to account for missing data using all available post-baseline data from Week 4 to Week 48 regardless of status on- or off-treatment used in the model (ITT analysis).
Time Frame: Baseline to Week 12
Population: Analysis was performed on ITT population which included all enrolled participants who had received at least one dose or partial dose of alirocumab. As pre-specified, efficacy analysis data were planned to be collected and analyzed for all doses combined (i.e. for combined population).
Measure: Least Squares Mean (Standard Error); unit: percent change
Groups:
- Alirocumab: All participants who received either 75 mg (BW <50 kg) or 150 mg (BW >=50 kg) alirocumab subcutaneously Q2W for 48 weeks.
Arm/Group | Alirocumab
Number analyzed (Participants) | 18
percent change | -4.1 (9.0)

2. Secondary Outcome: Percent Change From Baseline in Low-Density Lipoprotein Cholesterol at Week 12: On-treatment Analysis
Description: Adjusted LS means and standard errors were obtained from the MMRM model to account for missing data using all available post-baseline on-treatment data from Week 4 to Week 48 (on-treatment Analysis).
Time Frame: Baseline to Week 12
Population: Analysis was performed on ITT population. As pre-specified, efficacy analysis data were planned to be collected and analyzed for all doses combined (i.e. for combined population).
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Alirocumab
Number analyzed (Participants) | 18
percent change | -4.1 (9.0)

3. Secondary Outcome: Percent Change From Baseline in Low-Density Lipoprotein Cholesterol at Weeks 24 and 48: ITT Analysis/On-treatment Analysis
Description: Adjusted LS means and standard errors were obtained from the MMRM model to account for missing data using all available post-baseline data from Week 4 to Week 48 regardless of status on- or off-treatment used in the model (ITT analysis). Although separate analyses of all available data (ITT analysis) and only data collected within a defined time window (On-treatment analysis) were planned, if all values used in the ITT approach were within the on-treatment time window, the on-treatment analysis would be identical to the ITT analysis, thus the results would be identical and a single outcome measure presenting the results for both types of analysis would be provided.
Time Frame: Baseline to Weeks 24 and 48
Population: Analysis was performed on ITT population. As pre-specified, efficacy analysis data were planned to be collected and analyzed for all doses combined (i.e., for combined population).
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Alirocumab
Number analyzed (Participants) | 18
percent change
  Week 24 | -10.1 (7.6)
  Week 48 | 4.2 (12.8)

4. Secondary Outcome: Percent Change From Baseline in Apolipoprotein (Apo) B at Weeks 12, 24 and 48: ITT Analysis/On-treatment Analysis
Description: as for outcome 3
Time Frame: Baseline to Weeks 12, 24 and 48
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Alirocumab
Number analyzed (Participants) | 18
percent change
  Week 12 | -4.2 (6.8)
  Week 24 | -11.8 (6.1)
  Week 48 | 0.9 (10.4)

5. Secondary Outcome: Percent Change From Baseline in Non-High Density Lipoprotein Cholesterol (Non-HDL-C) at Weeks 12, 24 and 48 - ITT Analysis/On-treatment Analysis
Description: as for outcome 3
Time Frame: Baseline to Weeks 12, 24 and 48
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Alirocumab
Number analyzed (Participants) | 18
percent change
  Week 12 | -3.9 (8.3)
  Week 24 | -9.2 (7.3)
  Week 48 | 5.7 (13.1)

6. Secondary Outcome: Percent Change From Baseline in Total Cholesterol (Total-C) at Weeks 12, 24 and 48: ITT Analysis/On-treatment Analysis
Description: Adjusted LS means and standard errors were obtained from the MMRM model to account for missing data using all available post-baseline data from Weeks 4 to Week 48 regardless of status on- or off-treatment used in the model (ITT analysis). Although separate analyses of all available data (ITT analysis) and only data collected within a defined time window (On-treatment analysis) were planned, if all values used in the ITT approach were within the on-treatment time window, the on-treatment analysis would be identical to the ITT analysis, thus the results would be identical and a single outcome measure presenting the results for both types of analysis would be provided.
Time Frame: Baseline to Weeks 12, 24 and 48
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Alirocumab
Number analyzed (Participants) | 18
percent change
  Week 12 | -1.9 (7.2)
  Week 24 | -6.3 (6.5)
  Week 48 | 5.5 (10.7)

7. Secondary Outcome: Percent Change From Baseline in Lipoprotein a (Lp) (a) at Weeks 12, 24 and 48: ITT Analysis/On-treatment Analysis
Description: Adjusted means and standard errors were obtained from a multiple imputation approach followed by a robust regression model including all available post-baseline data from Week 4 to Week 48 regardless of status on-or off-treatment used in the model (ITT analysis). Although separate analyses of all available data (ITT analysis) and only data collected within a defined time window (On-treatment analysis) were planned, if all values used in the ITT approach were within the on-treatment time window, the on-treatment analysis would be identical to the ITT analysis, thus the results would be identical and a single outcome measure presenting the results for both types of analysis would be provided.
Time Frame: Baseline to Weeks 12, 24 and 48
Population: as for outcome 3
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Alirocumab
Number analyzed (Participants) | 18
percent change
  Week 12 | 7.4 (7.6)
  Week 24 | -5.2 (8.1)
  Week 48 | -6.4 (12.2)

8. Secondary Outcome: Percent Change From Baseline in High Density Lipoprotein Cholesterol (HDL-C) at Weeks 12, 24 and 48: ITT Analysis/On-treatment Analysis
Description: as for outcome 6
Time Frame: Baseline to Weeks 12, 24 and 48
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Alirocumab
Number analyzed (Participants) | 18
percent change
  Week 12 | 13.0 (5.9)
  Week 24 | 8.9 (4.4)
  Week 48 | 10.1 (5.5)

9. Secondary Outcome: Percent Change From Baseline in Fasting Triglycerides (TG) at Weeks 12, 24 and 48: ITT Analysis/On-treatment Analysis
Description: Adjusted means and standard errors were obtained from a multiple imputation approach followed by a robust regression model including all available post-baseline data from Week 4 to Week 48 regardless of status on- or off-treatment used in the model (ITT analysis). Although separate analyses of all available data (ITT analysis) and only data collected within a defined time window (On-treatment analysis) were planned, if all values used in the ITT approach were within the on-treatment time window, the on-treatment analysis would be identical to the ITT analysis, thus the results would be identical and a single outcome measure presenting the results for both types of analysis would be provided.
Time Frame: Baseline to Weeks 12, 24 and 48
Population: as for outcome 3
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Alirocumab
Number analyzed (Participants) | 18
percent change
  Week 12 | 2.8 (8.0)
  Week 24 | 5.2 (16.2)
  Week 48 | 10.0 (8.2)

10. Secondary Outcome: Percent Change From Baseline in Apolipoprotein A1 (Apo A1) at Weeks 12, 24 and 48: ITT Analysis/On-treatment Analysis
Description: Adjusted LS means and standard errors were obtained from the MMRM model to account for missing data using all available post-baseline data from Week 4 to 48 regardless of status on- or off-treatment used in the model (ITT analysis). Although separate analyses of all available data (ITT analysis) and only data collected within a defined time window (On-treatment analysis) were planned, if all values used in the ITT approach were within the on-treatment time window, the on-treatment analysis would be identical to the ITT analysis, thus the results would be identical and a single outcome measure presenting the results for both types of analysis would be provided.
Time Frame: Baseline to Weeks 12, 24 and 48
Population: Analysis was performed on ITT population. As pre-specified, efficacy analysis data was planned to be collected and analyzed for all doses combined (i.e., for combined population).
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Alirocumab
Number analyzed (Participants) | 18
percent change
  Week 12 | 11.3 (6.9)
  Week 24 | 14.6 (6.0)
  Week 48 | 11.3 (5.8)

11. Secondary Outcome: Percentage of Participants Reporting >=15 Percent (%) Reduction in LDL-C Level at Weeks 12, 24 and 48: ITT Analysis/On-treatment Analysis
Description: Adjusted Percentage were obtained from a multiple imputation approach for handling of missing data including all available post-baseline data from Week 4 to Week 48 regardless of status on- or off-treatment used in the model (ITT analysis). Although separate analyses of all available data (ITT analysis) and only data collected within a defined time window (On-treatment analysis) were planned, if all values used in the ITT approach were within the on-treatment time window, the on-treatment analysis would be identical to the ITT analysis, thus the results would be identical and a single outcome measure presenting the results for both types of analysis would be provided.
Time Frame: Baseline to Weeks 12, 24 and 48
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Alirocumab
Number analyzed (Participants) | 18
percentage of participants
  Week 12 | 50.0 [26.2 to 73.8]
  Week 24 | 50.0 [26.2 to 73.8]
  Week 48 | 39.0 [15.8 to 62.2]

12. Secondary Outcome: Absolute Change From Baseline in LDL-C Level at Weeks 12, 24 and 48: ITT Analysis/On-treatment Analysis
Description: as for outcome 3
Time Frame: Baseline to Weeks 12, 24 and 48
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Alirocumab
Number analyzed (Participants) | 18
mg/dL
  Week 12 | -33.4 (19.1)
  Week 24 | -43.0 (19.0)
  Week 48 | -15.0 (25.7)

13. Secondary Outcome: Number of Participants With Tanner Staging at Baseline, Weeks 12, 24 and 48
Description: Tanner stage defines physical measurements of development in children and adolescent based on external primary and secondary sex characteristics. Participants were evaluated for pubic hair distribution, breast development (only females) and genital development (only males), and classified in 3 categories as: Prepubescent (defined as a person just before start of the development of adult sexual characteristics), Pubescent (defined as a person at or approaching the age of puberty), Postpubescent (sexually mature or a person who has completed puberty).
Time Frame: Baseline, Weeks 12, 24 and 48
Population: Analysis was performed on safety population which included participants who had received at least one dose or partial dose of alirocumab. Here, 'number analyzed' = participants with available data for each specified category.
Measure: Count of Participants; unit: Participants
Arm/Group | Alirocumab 75 mg Q2W/up to 150 mg Q2W | Alirocumab 150 mg Q2W
Number analyzed (Participants) | 9 | 9
Participants
  Baseline: Prepubescent | 3 | 0
  Baseline: Pubescent | 6 | 9
  Baseline: Post-pubescent | 0 | 0
  Week 12: Prepubescent | 3 | 0
  Week 12: Pubescent | 6 | 8
  Week 12: Post-pubescent | 0 | 1
  Week 24: Prepubescent: number analyzed (Participants) | 8 | 9
  Week 24: Prepubescent | 2 | 0
  Week 24: Pubescent: number analyzed (Participants) | 8 | 9
  Week 24: Pubescent | 6 | 8
  Week 24: Post-pubescent: number analyzed (Participants) | 8 | 9
  Week 24: Post-pubescent | 0 | 1
  Week 48: Prepubescent: number analyzed (Participants) | 8 | 9
  Week 48: Prepubescent | 1 | 0
  Week 48: Pubescent: number analyzed (Participants) | 8 | 9
  Week 48: Pubescent | 7 | 7
  Week 48: Post-pubescent: number analyzed (Participants) | 8 | 9
  Week 48: Post-pubescent | 0 | 2

ADVERSE EVENTS:
Time Frame: All Adverse Events (AEs) were collected from signature of the informed consent form up to 56 weeks of the study regardless of seriousness or relationship to investigational product.
Description: Reported AEs and death were treatment-emergent AEs (TEAE) that developed/worsened, and death that occurred during TEAE period (the time from the first dose of alirocumab up to the last dose of alirocumab + 70 days [10 weeks]). Analysis was performed on safety population.
Arm/Group | Alirocumab 75 mg Q2W/up to 150 mg Q2W | Alirocumab 150 mg Q2W
All-Cause Mortality (participants affected / at risk) | 1/9 | 0/9
Serious Adverse Events (participants affected / at risk) | 1/9 | 0/9
Other Adverse Events (participants affected / at risk) | 8/9 | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Alirocumab 75 mg Q2W/up to 150 mg Q2W (N=9) | Alirocumab 150 mg Q2W (N=9)
Cardiac Failure (Cardiac disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Alirocumab 75 mg Q2W/up to 150 mg Q2W (N=9) | Alirocumab 150 mg Q2W (N=9)
Splenomegaly (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Aortic Valve Incompetence (Cardiac disorders) | 2 (2) | 1 (1)
Bicuspid Aortic Valve (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0)
Influenza Like Illness (General disorders) | 1 (1) | 0 (0)
Injection Site Pain (General disorders) | 1 (1) | 0 (0)
Injection Site Reaction (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Hepatomegaly (Hepatobiliary disorders) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 2 (2) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 2 (2)
Parvovirus B19 Infection (Infections and infestations) | 1 (1) | 0 (0)
Pharyngotonsillitis (Infections and infestations) | 1 (1) | 0 (0)
Upper Respiratory Tract Infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 0 (0)
Thermal Burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine Aminotransferase Increased (Investigations) | 0 (0) | 1 (1)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Tendon Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 2 (4) | 1 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea Paroxysmal Nocturnal (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dry Skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor supports publication of clinical trial results but may request that investigators temporarily delay or alter publications in order to protect proprietary information. The Sponsor may also require that the results of multicenter studies be published only in their entirety and not as individual site data.

DOCUMENTS (2):
  • Study Protocol (2018-09-11): https://cdn.clinicaltrials.gov/large-docs/15/NCT03510715/Prot_000.pdf
  • Statistical Analysis Plan (2020-01-27): https://cdn.clinicaltrials.gov/large-docs/15/NCT03510715/SAP_001.pdf